CLINICAL TRIAL: NCT04858971
Title: Effect of Dietary Advice Source on Perceptions of Information Accuracy and Intended Compliance
Brief Title: Survey of Diet and Health Beliefs
Status: Completed | Type: Observational
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GFHNRC337
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Dietary Guidelines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: No source will be indicated on information provided for review
  Interventions: Other: Perception of information source
- Government source: A government logo will be shown on information provided for review
  Interventions: Other: Perception of information source
- Medical source: A medical logo will be shown on information provided for review
  Interventions: Other: Perception of information source
- Social media source: A social media logo will be shown on information provided for review
  Interventions: Other: Perception of information source

INTERVENTIONS:
Other: Perception of information source — Participants will see the same health advice, with no source or one of three other sources indicated

SUMMARY:
The purpose of this research is to better understand people's health and diet knowledge, beliefs, attitudes, and practices. The researchers will use this information to implement better strategies to help Americans maintain more nutritious diets.

DETAILED DESCRIPTION:
The overall goal of this study is to determine whether there are differences in perceptions of healthy nutrition messages depending on from whom the message is coming. More specifically, the researchers aim to examine whether there are differences in how people perceive and intend to follow nutrition information that is coming from a variety of sources.

ELIGIBILITY:
Inclusion Criteria:

* US citizen
* have access to internet
* have an Amazon Mechanical Turk (MTurk) account

Exclusion Criteria:

* under 18 years of age
* no access to internet

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include American adults aged 18 and over. Minors, i.e., those under 18, will be excluded. To participate, people must have access to internet. Therefore, by default, those who do not have internet access will be excluded from this study. Due to the nature of this study, participants from all over the country will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Perception of health information | Baseline
  Participants will rate the extent to which they trust the source of health information (i.e., the makers of the flyer) on a 7-point Likert-type scale ranging from not at all (1) to completely (7).

CONTACTS AND LOCATIONS:
Overall Officials: Alese Nelson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center; James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT04858971/ICF_000.pdf